CLINICAL TRIAL: NCT03073018
Title: Prevention of Renal and Vascular Endstage Disease Intervention Trial
Acronym: PREVEND-IT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Collaborators: Dutch Kidney Foundation (Other); Netherlands Heart Foundation (Other)
Responsible Party: Principal Investigator, Prof. Wiek H. van Gilst, Principal Investigator, University Medical Center Groningen
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: METc 97/10/172
Record Dates: First submitted 2017-01-27; First posted 2017-03-08 (Actual); Last update posted 2017-03-10 (Actual); Status verified 2017-03

CONDITIONS: Microalbuminuria; Cardiovascular Diseases; Renal Disease
MeSH Terms: conditions — Cardiovascular Diseases; Kidney Diseases | interventions — Fosinopril; Pravastatin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- Fosinopril + Pravastatin (Experimental): Fosinopril (20 mg) + pravastatin (40 mg) once daily for 4 years
  Interventions: Drug: Fosinopril; Drug: Pravastatin
- Fosinopril + Placebo (Active Comparator): Fosinopril (20 mg) + pravastatin placebo once daily for 4 years
  Interventions: Drug: Fosinopril; Drug: Pravastatin Placebo
- Pravastatin + Placebo (Active Comparator): Pravastatin (40 mg) + fosinopril placebo once daily for 4 years
  Interventions: Drug: Pravastatin; Drug: Fosinopril Placebo
- Double Placebo (Placebo Comparator): Fosinopril placebo and pravastatin placebo once daily for 4 years
  Interventions: Drug: Fosinopril Placebo; Drug: Pravastatin Placebo

INTERVENTIONS:
Drug: Fosinopril — oral administration, capsules
  Other Names: Monopril
  Arms: Fosinopril + Placebo; Fosinopril + Pravastatin
Drug: Pravastatin — oral administration, capsules
  Other Names: Pravachol
  Arms: Fosinopril + Pravastatin; Pravastatin + Placebo
Drug: Fosinopril Placebo — oral administration, capsules
  Arms: Double Placebo; Pravastatin + Placebo
Drug: Pravastatin Placebo — oral administration, capsules
  Arms: Double Placebo; Fosinopril + Placebo

SUMMARY:
The Prevention of Renal and Vascular Endstage Disease Intervention Trial (PREVEND IT) was designed to determine whether intervention with the angiotensin-converting enzyme (ACE) inhibitor fosinopril and/or the hydroxymethylglutaryl coenzyme A reductase inhibitor pravastatin reduced cardiovascular and renal events in nonhypertensive, nonhypercholesterolemic subjects with microalbuminuria.

DETAILED DESCRIPTION:
This study describes the rationale, design, and baseline characteristics of a trial to determine whether treatment with fosinopril 20 mg/day and/or pravastatin 40 mg/ day will prevent cardiovascular and renal disease in nonhypertensive (RR <160/100 mm Hg and not using antihypertensive medication) and nonhypercholesterolemic (total cholesterol <8.0 or <5.0 mmol/L in case of previous myocardial infarction and not using lipid lowering medication) men and women with persistent microalbuminuria (urinary albumin excretion >10 mg/L once in an early morning spot urine and 15 to 300 mg/24-hour at least once in two 24-hour urine collections). The Prevention of REnal and Vascular ENdstage Disease Intervention Trial is a single-center, double-blind, randomized, placebo-controlled trial with a 2 x 2 factorial design. The 864 randomized subjects will be monitored for a minimum of 4 years and a maximum of 5 years. The primary efficacy parameter is defined as the combined incidence of all-cause mortality or hospital admission for documented (1) nonfatal myocardial infarction, (2) myocardial ischemia, (3) heart failure, (4) peripheral vascular disease, (5) cerebrovascular accident and/or (6) end-stage renal disease.

ELIGIBILITY:
Inclusion Criteria:

* Persistent microalbuminuria (urinary albumin excretion >10mg/L once in an early morning spot urine and 15 to 300 mg/24 hours at least once in two 24-hour urine samples)
* No hypertension (RR <160/100 mm Hg, no anti-hypertensive medication)
* No hypercholesterolemia (total cholesterol <8.0 or <5.0 mmol/L in case of previous myocardial infarction and not using lipid-lowering medication)

Exclusion Criteria:

* Creatinine clearance >60% of the normal age-adjusted value
* Serum potassium >5.5 mmol/L
* History of chronic liver disease
* Lactate dehydrogenase, aspartate-amino transferase or alanine-amino transferase >3 times the upper limit of normal
* Use of angiotensin-converting enzyme inhibitors or angiotensin II receptor antagonists
* Use of insulin
* Previously documented allergy or intolerance to study drugs
* Pregnant or nursing women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 864 (Actual)
Dates: Start 1998-04; Primary Completion 2003-06 (Actual); Study Completion 2003-11 (Actual)

PRIMARY OUTCOMES:
Combined incidence of all-cause mortality, MACE and/or end-stage renal disease | 4 years
  Combined incidence of all-cause mortality or hospital admission for documented (1) non-fatal myocardial infarction, (2) myocardial ischemia, (3) heart failure, (4) peripheral vascular disease, (5) cerebrovascular accident and/or (6) end-stage renal disease

SECONDARY OUTCOMES:
Incidence of all-cause mortality | 4 years
  Incidence of all-cause mortality
effect of treatment on microalbuminuria | 4 years
  albumin excretion mg/24 h
effect of treatment on LDL cholesterol | 4 years
  in mmol/L
effect of treatment on blood pressure | 4 years
  in mmHg
Incidence of hospital admission | 4 years
  Incidence of hospital admission for documented (1) non-fatal myocardial infarction, (2) myocardial ischemia, (3) heart failure, (4) peripheral vascular disease, (5) cerebrovascular accident and/or (6) end-stage renal disease

CONTACTS AND LOCATIONS:
Overall Officials: Wiek H van Gilst, PhD, Principal Investigator — University Medical Center Groningen

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Diercks GF, Janssen WM, van Boven AJ, Bak AA, de Jong PE, Crijns HJ, van Gilst WH. Rationale, design, and baseline characteristics of a trial of prevention of cardiovascular and renal disease with fosinopril and pravastatin in nonhypertensive, nonhypercholesterolemic subjects with microalbuminuria (the Prevention of REnal and Vascular ENdstage Disease Intervention Trial [PREVEND IT]). Am J Cardiol. 2000 Sep 15;86(6):635-8. doi: 10.1016/s0002-9149(00)01042-0. PMID 10980214
- [Background] Asselbergs FW, Diercks GF, Hillege HL, van Boven AJ, Janssen WM, Voors AA, de Zeeuw D, de Jong PE, van Veldhuisen DJ, van Gilst WH; Prevention of Renal and Vascular Endstage Disease Intervention Trial (PREVEND IT) Investigators. Effects of fosinopril and pravastatin on cardiovascular events in subjects with microalbuminuria. Circulation. 2004 Nov 2;110(18):2809-16. doi: 10.1161/01.CIR.0000146378.65439.7A. Epub 2004 Oct 18. PMID 15492322
- [Derived] Kofink D, Eppinga RN, van Gilst WH, Bakker SJL, Dullaart RPF, van der Harst P, Asselbergs FW. Statin Effects on Metabolic Profiles: Data From the PREVEND IT (Prevention of Renal and Vascular End-stage Disease Intervention Trial). Circ Cardiovasc Genet. 2017 Dec;10(6):e001759. doi: 10.1161/CIRCGENETICS.117.001759. PMID 29237679